CLINICAL TRIAL: NCT01077128
Title: [E S] A Greek, Post-marketing, Observational Study of the quAlity of Life in Patients With Psoriasis Treated With Adalimumab - GOAL Study
Brief Title: Greek Study of the Quality of Life in Patients With Psoriasis Treated With Adalimumab
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P11-984
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Results first posted 2014-02-21 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Psoriasis
Keywords: Psoriasis; Quality of life
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with psoriasis: All eligible patients with psoriasis treated with Adalimumab

SUMMARY:
Primary objective

* To evaluate the quality of life of Adalimumab treated patients over a period of 12 months

Secondary objectives

* To evaluate the long-term efficacy of Adalimumab in patients with moderate to severe chronic plaque psoriasis as prescribed by the dermatologists in day-to-day clinical practice and in accordance with the terms of the European marketing authorization.
* To evaluate changes in patients quality of life according to treatment response over a 12-month period
* To observe and assess the long term use and safety of Adalimumab as prescribed by the dermatologist in a normal clinical setting and in accordance with the terms of the European marketing authorization.

DETAILED DESCRIPTION:
The aim of this post-marketing observational study in adult patients with moderate to severe chronic plaque psoriasis is to obtain further data on patient's Quality of Life and assess the impact of Adalimumab treatment on patient's quality of life in conditions of day-to-day clinical practice in Greece. This study will further assess the relationship between clinical outcomes and patient-reported outcomes. As this is an observational study, Abbott will not provide the study drug. Humira will be prescribed according to the routine medical practice. The participating physicians are free to determine the appropriate therapy for each patient and make treatment choices as deemed clinically necessary.

The Dermatology Life Quality Index (DLQI) will be used to assess patient quality of life. The Dermatology Life Quality Index (DLQI) total scores range from 0 to 30, with 0 corresponding to the best quality of life and 30 to the worst. The Dermatology Life Quality Index (DLQI) has well-established reliability and validity as determined in several studies. Moreover, it is frequently used in clinical trials of psoriasis.

The physician's global assessment of disease severity (PGA) will be used to measure patients' disease status at the time of assessment. It is a 6-point scale measuring the degree of overall psoriatic lesion severity, and scores range from 0 (clear) to 5 (very severe).

Complementary, European Quality of Life-5 Dimensions health questionnaire (EQ5D) will be used as a measure of health outcome. This is applicable to a wide range of health conditions and treatments and it provides a simple descriptive profile and a single index value for health status. Health economic data will be collected by using European Quality of Life-5 Dimensions health questionnaire (EQ5D) questionnaire and data regarding patients hospitalisation due to psoriasis. Hospitalisation data will be collected 6 months before the period and throughout the observation period.

Moreover, this study will observe the current medical practice in prescribing Adalimumab in Greece and more detailed data on prescription behavior will be collected. Guidelines have been developed in order to ensure that the new class of therapy (biologic agents) is introduced in a systematic and planned way to achieve the greatest possible benefit to people with psoriasis and to facilitate safe and effective prescribing. However, many issues are not fully addressed, such as recommendation regarding the amount of time for wash out of previous antipsoriatic drugs and combination therapies. Such issues remain at the discretion of the healthcare professional. Since this is an observational study the patient will be treated in accordance with the physician's usual and customary medical practice. Thus, the following information regarding the use of Adalimumab will be collected

* the previous systemic treatment history will be recorded including previous biological therapies that patient received, if any,
* wash out periods prior to initiating Adalimumab therapy, if any
* reasons for stopping previous treatment,
* combination of Adalimumab with other topical or systemic antipsoriatic agents, if applicable

Furthermore, demographic data of patients suffering from psoriasis in Greece will be collected (age, gender, ethnicity) and disease data such as duration of the disease, involvement of nails or joints, geographic distribution of the disease in Greece will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe chronic plaque psoriasis who are newly prescribed Humira (adalimumab) therapy (have never been treated with adalimumab before) and for whom the treating physician has made the decision that they are eligible for treatment with adalimumab in accordance with the terms of the local marketing authorization
* Patients with moderate to severe chronic plaque psoriasis for whom Adalimumab is indicated and has been prescribed according to the current approved local SPC as long as the first administration of adalimumab is not older than two months and they have not had dose interruptions since the initiation of adalimumab, and the Investigator can provide all the needed source documentation including a completed DLQI questionnaire at the start of Adalimumab treatment.
* Patient age ≥ 18
* Patient is willing to consent to data being collected and provided to Abbott

Exclusion Criteria:

* Patients who meet contraindications as outlined in the latest version of the local approved SPC
* Patients who participate in another clinical/observational study
* Patients who are not willing to sign an Informed Consent Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Adalimumab according to routine medical practice from hospital and private physicians.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athina Katsavou, MD, Study Chair — AbbVie Pharmaceuticals S.A.
Locations (61):
- Greece (61):
  - Site Reference ID/Investigator# 43746, Agrinio
  - Site Reference ID/Investigator# 30197, Amaliáda
  - Site Reference ID/Investigator# 30039, Argos
  - Site Reference ID/Investigator# 29903, Argyroúpoli
  - Site Reference ID/Investigator# 29819, Athens
  - Site Reference ID/Investigator# 29949, Athens
  - Site Reference ID/Investigator# 30804, Athens
  - Site Reference ID/Investigator# 30806, Athens
  - Site Reference ID/Investigator# 38324, Athens
  - Site Reference ID/Investigator# 22385, Athens
  - Site Reference ID/Investigator# 29826, Athens
  - Site Reference ID/Investigator# 29966, Athens
  - Site Reference ID/Investigator# 29991, Athens
  - Site Reference ID/Investigator# 30106, Athens
  - Site Reference ID/Investigator# 30107, Athens
  - Site Reference ID/Investigator# 30181, Athens
  - Site Reference ID/Investigator# 30470, Athens
  - Site Reference ID/Investigator# 30086, Chania, Crete
  - Site Reference ID/Investigator# 43744, Chania, Crete
  - Site Reference ID/Investigator# 30794, Crete
  - Site Reference ID/Investigator# 29937, Crete
  - Site Reference ID/Investigator# 29959, Crete
  - Site Reference ID/Investigator# 29969, Crete
  - Site Reference ID/Investigator# 38334, Drama
  - Site Reference ID/Investigator# 30801, Florina
  - Site Reference ID/Investigator# 29919, Giannitsá
  - Site Reference ID/Investigator# 30202, Giannitsá
  - Site Reference ID/Investigator# 29970, Glyfada
  - Site Reference ID/Investigator# 30013, Glyfada
  - Site Reference ID/Investigator# 29823, Glyfada
  - Site Reference ID/Investigator# 30193, Halandri
  - Site Reference ID/Investigator# 30083, Kalamaria
  - Site Reference ID/Investigator# 30143, Kallithea
  - Site Reference ID/Investigator# 47262, Katerini
  - Site Reference ID/Investigator# 38329, Keratsini
  - Site Reference ID/Investigator# 30108, Kolonaki
  - Site Reference ID/Investigator# 30009, Kosmos
  - Site Reference ID/Investigator# 38323, Larissa
  - Site Reference ID/Investigator# 38340, Larissa
  - Site Reference ID/Investigator# 29822, Livadeia
  - Site Reference ID/Investigator# 30180, Makri
  - Site Reference ID/Investigator# 29834, Mytilene
  - Site Reference ID/Investigator# 30469, Mytilene
  - Site Reference ID/Investigator# 38326, N.Heraklion
  - Site Reference ID/Investigator# 30032, Neapoli
  - Site Reference ID/Investigator# 30104, Pagkráti
  - Site Reference ID/Investigator# 29817, Pátrai
  - Site Reference ID/Investigator# 29967, Peiraius
  - Site Reference ID/Investigator# 38327, Peristeri
  - Site Reference ID/Investigator# 30109, Petralona
  - Site Reference ID/Investigator# 29824, Smyrni
  - Site Reference ID/Investigator# 38325, Thessaloniki
  - Site Reference ID/Investigator# 30769, Thessaloniki
  - Site Reference ID/Investigator# 30170, Thessaloniki
  - Site Reference ID/Investigator# 38331, Thessaloniki
  - Site Reference ID/Investigator# 38332, Thessaloniki
  - Site Reference ID/Investigator# 38333, Thessaloniki
  - Site Reference ID/Investigator# 38335, Thessaloniki
  - Site Reference ID/Investigator# 38337, Thessaloniki
  - Site Reference ID/Investigator# 30203, Vári
  - Site Reference ID/Investigator# 29921, Volos

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Psoriasis
Started | 500
Completed | 433
Not Completed | 67
Not completed — Adverse Event | 8
Not completed — Lack of Efficacy | 1
Not completed — Disease exacerbation | 1
Not completed — Adverse event and consent withdrawal | 1
Not completed — Adverse event and disease exacerbation | 1
Not completed — Lack of efficacy/disease exacerbation | 1
Not completed — Other | 54

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Psoriasis
Number analyzed (Participants) | 500
Age, Customized [Number; unit: participants]
  >=18 years | 500
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190
  Male | 310
Region of Enrollment [Number; unit: participants]
  Greece | 500
Regions of Greece [Number; unit: Participants]
  Attica | 266
  Central Macedonia | 71
  Crete | 41
  West Greece | 33
  East Macedonia and Thrace | 20
  Thessaly | 18
  Central Greece | 16
  Peloponnese | 16
  North Aegean | 8
  Ionian Islands | 4
  West Macedonia | 3
  South Aegean | 2
  Epirus | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change of Dermatology Life Quality Index (DLQI) Scores
Description: DLQI (Dermatology Life Quality Index) assesses symptoms and impacts of dermatologic diseases on quality of life. DLQI scores range from 0 to 30, with a higher score indicating a more impaired quality of life.
Time Frame: 12-month period, (Month 0, Month 1, Month 4, Month 8, Month 12)
Population: Participants with available data at each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Patients With Psoriasis- Month 1; Patients With Psoriasis- Month 4; Patients With Psoriasis- Month 8; Patients With Psoriasis- Month 12: All eligible patients with psoriasis treated with Adalimumab
Arm/Group | Patients With Psoriasis- Month 1 | Patients With Psoriasis- Month 4 | Patients With Psoriasis- Month 8 | Patients With Psoriasis- Month 12
Number analyzed (Participants) | 491 | 467 | 443 | 432
units on a scale | 4.9 (6.3) | 9.3 (7.3) | 11.3 (7.8) | 12.1 (7.8)

2. Secondary Outcome: Percentage of Patients Who Experienced an Improvement in Disease Severity as Determined by the Physician's Global Assessment of Disease Severity (PGA) Scores
Description: The Physician's Global Assessment of disease severity (PGA) was used to measure participants' disease status at the time of assessment. This tool is a horizontal visual analogue 6-point scale measuring the degree of overall psoriatic lesion severity, and scores range from 0 (clear) to 5 (very severe). The percentage of patients who showed an improvement from baseline in their PGA scores was recorded.
Time Frame: 12-month period (Month 0, Month 1, Month 4, Month 8, Month 12)
Population: Participants with available data at each time point
Measure: Number; unit: Percentage of patients improving
Arm/Group | Patients With Psoriasis- Month 1 | Patients With Psoriasis- Month 4 | Patients With Psoriasis- Month 8 | Patients With Psoriasis- Month 12
Number analyzed (Participants) | 491 | 470 | 445 | 433
Percentage of patients improving | 66.2 | 95.1 | 97.5 | 97.9

3. Secondary Outcome: Mean Change in the Dermatology Life Quality Index (DLQI) Score by Physician's Global Assessment of Disease Severity (PGA) Response Groups and by Geographical Region
Description: The average change in the Dermatology Life Quality Index (DLQI) score during the 12-month study was analyzed by the Physician's Global Assessment of disease severity (PGA) response and also by geographical location of study participants. DLQI scores range from 0 to 30, with a higher score indicating a more impaired quality of life. . In this table, a higher number means a greater improvement in the participants' quality of life.
Time Frame: 12-month period (Month 0, Month 1, Month 4, Month 8, Month 12)
Population: Participants with available data at each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- DLQI Score Change by PGA Response Group- Month 1; DLQI Score Change by PGA Response Group- Month 4; DLQI Score Change by PGA Response Group- Month 8; DLQI Score Change by PGA Response Group- Month 12; DLQI Score Change Baseline to Month 12- Attica; DLQI Score Change Baseline to Month 12- Central Greece; DLQI Score Change Baseline to Month 12- Central Macedonia; DLQI Score Change Baseline to Month 12- Crete; DLQI Score Change Baseline to Month 12- East Macedonia/Thrace; DLQI Score Change Baseline to Month 12- Epirus; DLQI Score Change Baseline to Month 12- Ionian Islands; DLQI Score Change Baseline to Month 12- North Aegean; DLQI Score Change Baseline to Month 12- Peloponnese; DLQI Score Change Baseline to Month 12- South Aegean; DLQI Score Change Baseline to Month 12- Thessaly; DLQI Score Change Baseline to Month 12- West Greece; DLQI Score Change Baseline to Month 12- West Macedonia: All eligible patients with psoriasis treated with Adalimumab
Arm/Group | DLQI Score Change by PGA Response Group- Month 1 | DLQI Score Change by PGA Response Group- Month 4 | DLQI Score Change by PGA Response Group- Month 8 | DLQI Score Change by PGA Response Group- Month 12 | DLQI Score Change Baseline to Month 12- Attica | DLQI Score Change Baseline to Month 12- Central Greece | DLQI Score Change Baseline to Month 12- Central Macedonia | DLQI Score Change Baseline to Month 12- Crete | DLQI Score Change Baseline to Month 12- East Macedonia/Thrace | DLQI Score Change Baseline to Month 12- Epirus | DLQI Score Change Baseline to Month 12- Ionian Islands | DLQI Score Change Baseline to Month 12- North Aegean | DLQI Score Change Baseline to Month 12- Peloponnese | DLQI Score Change Baseline to Month 12- South Aegean | DLQI Score Change Baseline to Month 12- Thessaly | DLQI Score Change Baseline to Month 12- West Greece | DLQI Score Change Baseline to Month 12- West Macedonia
Number analyzed (Participants) | 325 | 444 | 433 | 423 | 237 | 16 | 65 | 34 | 20 | 2 | 1 | 7 | 10 | 2 | 15 | 21 | 2
units on a scale | 6.3 (6.5) | 9.6 (7.1) | 11.5 (7.7) | 12.3 (7.8) | 12.9 (8.5) | 14.9 (7.2) | 12.3 (6.4) | 11.2 (6.7) | 10.6 (6.1) | 2.0 (0.0) | 19.0 | 11.0 (7.7) | 6.8 (4.7) | 15.0 (4.2) | 9.5 (7.7) | 8.7 (7.2) | 12.5 (2.1)

4. Secondary Outcome: Percentage of Patients Reporting "No Problem" on the European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D)
Description: EQ-5D (European Quality of Life - 5 Dimensions Questionnaire) is a standardized instrument for use as a measure of health outcome.
  It has two components:
  1. the EQ-5D descriptive system (i.e., the EQ-5D Index Score, comprised of five items), and
  2. the EQ-5D VAS. The EQ-5D Index Score has five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Patients reported either "problem" or "no problem" with each of the five dimensions of health. The EQ-5D VAS is a 20-cm scale with endpoints labeled "best imaginable health" and "worst imaginable health" anchored at 100 and 0, respectively.
Time Frame: 12-month period (Month 0, Month 1, Month 4, Month 8, Month 12)
Population: Participants with available data at each time point
Measure: Number; unit: Percentage of patients with no problem
Groups:
- EQ5D- Mobility- Baseline; EQ5D- Mobility- Month 1; EQ5D- Mobility- Month 4; EQ5D- Mobility- Month 8; EQ5D- Mobility- Month 12; EQ5D- Self-care- Baseline; EQ5D- Self-care- Month 1; EQ5D- Self-care- Month 4; EQ5D- Self-care- Month 8; EQ5D- Self-care- Month 12; EQ5D- Usual Activities- Baseline; EQ5D- Usual Activities- Month 1; EQ5D- Usual Activities- Month 4; EQ5D- Usual Activities- Month 8; EQ5D- Usual Activities- Month 12; EQ5D- Pain/Discomfort- Baseline; EQ5D- Pain/Discomfort- Month 1; EQ5D- Pain/Discomfort- Month 4; EQ5D- Pain/Discomfort- Month 8; EQ5D- Pain/Discomfort- Month 12; EQ5D- Anxiety/Depression- Baseline; EQ5D- Anxiety/Depression- Month 1; EQ5D- Anxiety/Depression- Month 4; EQ5D- Anxiety/Depression- Month 8; EQ5D- Anxiety/Depression- Month 12: All eligible patients with psoriasis treated with Adalimumab
Arm/Group | EQ5D- Mobility- Baseline | EQ5D- Mobility- Month 1 | EQ5D- Mobility- Month 4 | EQ5D- Mobility- Month 8 | EQ5D- Mobility- Month 12 | EQ5D- Self-care- Baseline | EQ5D- Self-care- Month 1 | EQ5D- Self-care- Month 4 | EQ5D- Self-care- Month 8 | EQ5D- Self-care- Month 12 | EQ5D- Usual Activities- Baseline | EQ5D- Usual Activities- Month 1 | EQ5D- Usual Activities- Month 4 | EQ5D- Usual Activities- Month 8 | EQ5D- Usual Activities- Month 12 | EQ5D- Pain/Discomfort- Baseline | EQ5D- Pain/Discomfort- Month 1 | EQ5D- Pain/Discomfort- Month 4 | EQ5D- Pain/Discomfort- Month 8 | EQ5D- Pain/Discomfort- Month 12 | EQ5D- Anxiety/Depression- Baseline | EQ5D- Anxiety/Depression- Month 1 | EQ5D- Anxiety/Depression- Month 4 | EQ5D- Anxiety/Depression- Month 8 | EQ5D- Anxiety/Depression- Month 12
Number analyzed (Participants) | 500 | 491 | 469 | 445 | 433 | 500 | 491 | 469 | 445 | 432 | 500 | 491 | 468 | 445 | 433 | 500 | 491 | 469 | 445 | 431 | 500 | 491 | 467 | 445 | 433
Percentage of patients with no problem | 74.6 | 66.2 | 90.2 | 91.5 | 90.8 | 81.2 | 84.3 | 92.1 | 95.3 | 94.2 | 66.2 | 77.8 | 90.2 | 92.1 | 94.5 | 56.2 | 73.1 | 87.2 | 90.3 | 93.3 | 20.8 | 36.9 | 53.7 | 67.6 | 73.0

5. Secondary Outcome: Mean Change From Baseline of European Quality of Life-5 Dimensions Health Questionnaire (EQ-5D) Visual Analogue Scale (VAS) Scores
Description: EQ-5D (European Quality of Life - 5 Dimensions Questionnaire) is a standardized instrument for use as a measure of health outcome.
  It has two components:
  1. the EQ-5D descriptive system (i.e., the EQ-5D Index Score, comprised of five items), and
  2. the EQ-5D VAS. EQ-5D Index Score has five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Patients reported either "problem" or "no problem" with each of the five dimensions of health. The EQ-5D VAS is a 20-cm scale with endpoints labeled "best imaginable health" and "worst imaginable health" anchored at 100 and 0, respectively.
Time Frame: 12-month period (Month 0, Month 1, Month 4, Month 8, Month 12)
Population: Participants with available data at each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- EQ-5D VAS- Mean Change From Baseline-Month 1; EQ-5D VAS- Mean Change From Baseline-Month 4; EQ-5D VAS- Mean Change From Baseline-Month 8; EQ-5D VAS- Mean Change From Baseline-Month 12: All eligible patients with psoriasis treated with Adalimumab
Arm/Group | EQ-5D VAS- Mean Change From Baseline-Month 1 | EQ-5D VAS- Mean Change From Baseline-Month 4 | EQ-5D VAS- Mean Change From Baseline-Month 8 | EQ-5D VAS- Mean Change From Baseline-Month 12
Number analyzed (Participants) | 491 | 470 | 445 | 433
units on a scale | 12.5 (15.8) | 25.9 (20.5) | 31.8 (23.3) | 35.9 (22.4)

6. Secondary Outcome: Assessment of Long Term Use and Safety of Adalimumab as Prescribed by the Dermatologist in a Normal Clinical Setting and in Accordance With the Terms of the European Marketing Authorization
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant, which did not necessarily have a causal relationship with their treatment. Any worsening of a pre-existing condition or illness was considered an adverse event.
Time Frame: 12-month period (Month 0, Month 1, Month 4, Month 8, Month 12)
Measure: Number; unit: Participants
Groups:
- Patients With Psoriasis: All eligible patients with psoriasis treated with Adalimumab were followed for the long term use and safety of Adalimumab. For more detailed information, please see the Adverse Events section.
Arm/Group | Patients With Psoriasis
Number analyzed (Participants) | 500
Participants | 500

ADVERSE EVENTS:
Time Frame: Data on adverse events were collected from study enrollment (Month 0) through Month 12.
Arm/Group | Patients With Psoriasis
Serious Adverse Events (participants affected / at risk) | 11/500
Other Adverse Events (participants affected / at risk) | 0/500
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Psoriasis (N=500)
Dysarthria (Nervous system disorders) | 1
Extradural haematoma (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Paresis (Nervous system disorders) | 1
Spinal cord ischaemia (Nervous system disorders) | 1
Spinal haematoma (Nervous system disorders) | 1
Eosinophilia (Blood and lymphatic system disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1
Asthenia (General disorders) | 2
Pyrexia (General disorders) | 2
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Oedema, peripheral (General disorders) | 1
Muscle contractions involuntary (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Ischaemic stroke (Vascular disorders) | 2
Transient ischaemic attack (Vascular disorders) | 1
Thyroiditis acute (Endocrine disorders) | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Electromyogram abnormal (Investigations) | 1
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Abortion induced (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.